CLINICAL TRIAL: NCT04190641
Title: Clinical Investigation to Evaluate the Direct Visualization Performances of Ambu® aScope™ 4 Cysto and aView™ Urologia for Examination of the Lower Urinary Tract
Brief Title: Single-use Cystoscope System for Direct Visualization of the Urethra and Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ambu A/S (Industry)
Collaborators: QserveCRO (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIS-013
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2020-08

CONDITIONS: Cystoscope; Bladder Cancer; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Urinary Bladder Neoplasms; Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: A non-randomized confirmatory study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Flexible cystoscopy (Other): Visualization of the urethra and bladder with the Ambu® aScope™ 4 Cysto and aView™ Urologia
  Interventions: Device: Ambu aScope 4 Cysto and aView Urologia

INTERVENTIONS:
Device: Ambu aScope 4 Cysto and aView Urologia — Visualization of the urethra and the bladder

SUMMARY:
In this study, the new aScope 4 Cysto is used to see how well it visualizes the lower urinary tract, and if this new flexible cystoscope performs as well as other routinely used cystoscopes. This study will be done in patients who have been diagnosed with bladder lesions and who will undergo surgery via the urethra to remove these lesions. The surgery is done under general anesthesia. After being brought under anesthesia and before removal of the lesion(s), the new flexible cystoscope is tested. The cystoscope will be used to visualize the urethra and bladder. Data will be collected on the number of the lesions that can be seen using the new cystoscope. During the planned surgery a resectoscope or rigid cystoscope will be used to confirm the number of lesions. The data will be used to show how well the cystoscope visualizes the lesions in comparison with routinely used cystoscopes. It will give information on how well the structures of the urinary tract and bladder can be viewed including any abnormalities that are present.Data will also be collected on the handling of the cystoscope: how well the cystoscope moves into the lower urinary tract, and how well it can be navigated through the lower urinary tract.

DETAILED DESCRIPTION:
Clinical Phase: pre-CE study

Design: A non-randomized confirmatory study on the visualization performance of the Ambu® aScope™ 4 Cysto and aView™ Urologia in 42 fully evaluable, adults subjects aimed at identification of known pathological findings (papillary bladder or small resectable lesion) detected with Ambu® aScope™ 4 Cysto and aView™ Urologia and subsequently during a repeat procedure using a reusable rigid scope or resectoscope at the time of planned transurethral resection of bladder tumours (TURBT).

Population: Adult subjects (≥ 18 years) in the OR undergoing planned transurethral resection of bladder tumors TURBT

Planned sample size: A total of 42 patients will result in a maximum (if the true proportion is 50 %) width of the two-sided 95 % confidence interval for the binary variable "Confirmed" to be 15%. This width is considered to be useful in the interpretations of the results from this investigation.

Study duration: Screening, procedure and follow-up will take 15 days maximum

Follow-up duration: Follow-up immediately after procedure

Investigational Device: Ambu® aScope™ 4 Cysto and aView™ Urologia Pre-CE, single use cystoscope.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign the informed consent
* Adults (males and females), ≥18 years of age or older
* Able to undergo routine cystoscopy
* Patients diagnosed with papillary bladder or small resectable lesion where transurethral resection of the tumour/lesion is planned

Exclusion Criteria:

* History of prior bladder/urethral reconstructive surgery
* Presence of symptomatic urinary tract infection (UTI)
* Known unpassable urethral stricture
* Unable to read and/or understand the study requirements
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-07-06 (Actual)

PRIMARY OUTCOMES:
performance of Ambu® aScope™ 4 Cysto and aView™ Urologia | follow up immediately after procedure
  The performance level of Ambu® aScope™ 4 Cysto and aView™ Urologia, compared to current standard practice with re-usable cystoscopes, is defined as proportion of patients with one or more papillary bladder lesion or small resectable lesion (diagnosed a maximum of one month prior to resection) detected with the Ambu® aScope™ 4 Cysto and aView™ Urologia (prior to planned transurethral resection of bladder tumors (TURBT)) and confirmed with the rigid cystoscope during TURBT.

SECONDARY OUTCOMES:
Safety of Ambu® aScope™ 4 Cysto and aView™ Urologia | follow up immediately after procedure
  Evaluate the safety of Ambu® aScope™ 4 Cysto and aView™ Urologia for direct visualization of the urethra and bladder by assessing the adverse events during and immediately after the flexible cystoscopy with Ambu® aScope™ 4 Cysto and aView™ Urologia, prior to start of TURBT
Investigator performance | follow up immediately after procedure
  Measure of the overall performance by using a 5-point Likert scale with a minimum of one (=worst possible) to maximum of five (=best possible), to be completed by the investigator that performed the cystoscopy.
Procedure time | follow up immediately after procedure
  Measure of the overall procedure time

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No